CLINICAL TRIAL: NCT05092997
Title: Interventions for Improved Post-partum ART Continuation and HIV Testing of Male Partners of Women in PMTCT B+ in Uganda (Kingasa Study)
Brief Title: Kingasa Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Harvard University (Other)
Responsible Party: Principal Investigator, Connie Celum, Professor of Global Health, Medicine, and Epidemiology, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00009286; R01MH113434 (NIH)
Record Dates: First submitted 2021-07-26; First posted 2021-10-26 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: HIV; Linkage to Care; PMTCT; PrEP; ART Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Female SOC/Male SOC arm (No Intervention): Women will be provided the standard of care invitation letter for male partners for fast-track visit for HIV testing and laboratory HIV testing at enrollment and every 6 months until 6 months postpartum,
- Female intervention/Male SOC arm (Active Comparator): Women will be provided the standard of care invitation letter for male partners for fast-track visit for HIV testing and POC VL tests for women at enrollment, delivery, and 6 months post-partum;
  Interventions: Diagnostic Test: POC viral load testing
- Female SOC/Male intervention arm (Active Comparator): Women will be provided an invitation letter for male partners for wellness visits and laboratory-based HIV VL testing for women at enrollment, delivery, and 6 months post-partum;
  Interventions: Other: Wellness visit services for male partners
- Female intervention/male intervention arm (Active Comparator): Women will be provided an invitation letter for male partners invitation letter for male partners for wellness visits and POC viral load testing for women at enrollment, delivery, and 6 months post-partum.
  Interventions: Diagnostic Test: POC viral load testing; Other: Wellness visit services for male partners

INTERVENTIONS:
Diagnostic Test: POC viral load testing — POC viral load testing- women randomized to have POC VL at enrollment, delivery and 6 months post-partum, will have a finger prick to obtain whole blood for the Cepheid Xpert HIV-1 RNA cartridge on the Xpert IV machine with results in 90 minutes. Women who are randomized to POC VL who have VL >200 c/ml will receive additional adherence counseling, following the STREAM protocol, [26] to address the challenges that they are having with ART use. At the delivery visit, infants of women in the POC VL arm will also have viral load testing done.
  Arms: Female intervention/Male SOC arm; Female intervention/male intervention arm
Other: Wellness visit services for male partners — Wellness visits for men- additional prevention services for men randomized to the intervention arm, including dual syphilis and HIV testing, blood pressure, visual acuity screening, and COVID-19 screening as part of wellness
  Arms: Female SOC/Male intervention arm; Female intervention/male intervention arm

SUMMARY:
In the Kingasa study, the investigators will use a factorial design in order to evaluate both an intervention to increase male partner HIV testing and an intervention for pregnant and postpartum women living with HIV to provide real-time HIV VL load and ART adherence counseling. Specifically, the investigators will evaluate a) whether invitations to wellness visits increase the proportion of male partners who test for HIV and b) whether POC HIV VL tests increase viral suppression among pregnant and postpartum women living with HIV. The research team will also assess the impact of providing male counselor phone call follow-up to men in the wellness visit arm to encourage linkage to HIV care and prevention after HIV testing. Women will be randomized 1:1:1:1 to receive a) standard of care interventions with an invitation letter for male partners for fast-track visit for HIV testing and laboratory HIV testing for women at enrollment and every 6 months until 12 months postpartum, b) invitation letter for male partners for fast track visit for HIV testing and POC VL tests for women at enrollment and every 6 months until 12 months postpartum; c) invitation letter to male partners for wellness visits and laboratory-based HIV VL testing for women at enrollment and every 6 months until 12 months postpartum; and d) invitation letter to male partners for wellness visits and POC viral load testing for women at enrollment and every 6 months until 12 months post-partum. Women who are randomized to receive POC VL will receive same-day ART adherence counseling and those randomized to receive lab-based VL will receive VL results at their next visit with ART adherence counseling based on their VL results.

DETAILED DESCRIPTION:
In the Kingasa study, the investigators will use a factorial design in order to evaluate both an intervention to increase male partner HIV testing and an intervention for pregnant and postpartum women living with HIV to provide real-time HIV VL load and ART adherence counseling. Specifically, the investigators will evaluate a) whether invitations to wellness visits increase the proportion of male partners who test for HIV and b) whether POC HIV VL tests increase viral suppression among pregnant and postpartum women living with HIV. The research team will also assess the impact of providing male counselor phone call follow-up to men in the wellness visit arm to encourage linkage to HIV care and prevention after HIV testing. Women will be randomized 1:1:1:1 to receive a) standard of care interventions with an invitation letter for male partners for fast-track visit for HIV testing and laboratory HIV testing for women at enrollment and every 6 months until 12 months postpartum, b) invitation letter for male partners for fast track visit for HIV testing and POC VL tests for women at enrollment and every 6 months until 12 months postpartum; c) invitation letter to male partners for wellness visits and laboratory-based HIV VL testing for women at enrollment and every 6 months until 12 months postpartum; and d) invitation letter to male partners for wellness visits and POC viral load testing for women at enrollment and every 6 months until 12 months post-partum. Women who are randomized to receive POC VL will receive same day ART adherence counseling and those randomized to receive lab based VL will receive VL results at their next visit with ART adherence counseling based on their VL results.

Women in both arms will receive counseling to minimize social harms associated with status disclosure and HIV testing, and additional counseling and referral to social support services when social harms occur. Based on the current Ugandan MOH guidelines to offer HIVST to both HIV-positive and HIV-negative pregnant women in ANC clinics, women in both arms will be provided an HIVST to give to their partner if they choose. They will be trained in the use and interpretation of the HIVST and be given information about HIV testing and prevention and care services, which she will give to her partner.

This study has been designed to address the gap in male partner engagement by using innovative methods to link men to HIV testing, prevention and care, and thus PMTCT outcomes for women.

ELIGIBILITY:
Inclusion Criteria for women:

* Age ≥18 or 14-17 years if an emancipated minor (pregnant or have a child)
* Currently pregnant
* Not currently enrolled in an HIV treatment study
* Male partner not known to be HIV-positive or has not tested in the past 3 months
* Able and willing to provide written informed consent
* Able and willing to provide adequate locator information for study retention purposes
* Screening negative for any indication of intimate partner violence or social harm

Inclusion Criteria for men:

- female partner enrolled in Kingasa pilot study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Male partner HIV testing | 6 months from female partner enrollment
  To determine the proportion of male partners of pregnant HIV-positive women who test for HIV at the clinic, based on invitation to a wellness visit (dual syphilis and HIV rapid test, blood pressure, visual acuity screening and COVID symptom screening, and if available, PCR testing for those with symptoms) compared to the standard of care (standard of care invitation letter for HIV fast track testing at the clinic).
Viral suppression | 6 months post-partum
  To compare viral suppression (defined as less than 50 copies/mL) at 6 months post-partum among women in the intervention arm (receiving POC viral load testing and same-day ART adherence support) to women in the control arm (receiving stand of care lab-based HIV VL testing).
Male partner linkage | 6 months from female partner enrollment
  To assess the proportion of HIV-negative male partners who initiate PrEP and HIV positive men who initiate ART among male partners who test for HIV and are provided male counselor phone follow up or who receive standard of care.
Acceptability evaluation | One time point at 3 months post-partum for women, and one time point at 3 months post enrollment for men
  To evaluate acceptability and preferences for HIV testing and other health services among 15 pregnant women and 15 male partners using qualitative in-depth interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Disease Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ware NC, Wyatt MA, Nakyanzi A, Naddunga F, Pisarski EE, Kyomugisha J, Birungi JE, Bulterys MA, Kamusiime B, Nalumansi A, Kasiita V, Mujugira A, Celum CL. POC Viral Load Testing in an Antenatal Clinic Setting for Ugandan Pregnant Women Living with HIV: An Implementation Process Analysis. Discov Health Syst. 2024;3:44. doi: 10.1007/s44250-024-00103-8. Epub 2024 Jun 26. PMID 39896214

DOCUMENTS (1):
  • Study Protocol (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05092997/Prot_000.pdf